CLINICAL TRIAL: NCT01456364
Title: Prospective, Randomized Study of the Platelet Inhibitory Efficacy of Ticagrelor Versus Prasugrel in Clopidogrel Low Responders After Percutaneous Coronary Intervention
Brief Title: Intracoronary Stenting and Antithrombotic Regimen: ADjusting Antiplatelet Treatment in PatienTs Based on Platelet Function Testing
Acronym: ISAR ADAPT PF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GE-DHM A01811
Record Dates: First submitted 2011-10-18; First posted 2011-10-20 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Coronary Heart Disease
Keywords: clopidogrel low response; ticagrelor; prasugrel; platelet aggregation
MeSH Terms: conditions — Coronary Disease | interventions — Ticagrelor; Prasugrel Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ticagrelor (Active Comparator): A loading dose of 180 mg of ticagrelor is administered followed by 90 mg maintenance doses twice daily
  Interventions: Drug: Ticagrelor
- Prasugrel (Active Comparator): A prasugrel loading dose of 60 mg is administered followed by a 10 mg per day maintenance dose for patients < 75 years or a 5 mg maintenance dose per day for patients >= 75 years
  Interventions: Drug: Prasugrel

INTERVENTIONS:
Drug: Ticagrelor — A loading dose of 180 mg of ticagrelor is administered followed by 90 mg maintenance doses twice daily
  Arms: Ticagrelor
Drug: Prasugrel — A prasugrel loading dose of 60 mg is administered followed by a 10 mg per day maintenance dose for patients < 75 years or a 5 mg maintenance dose per day for patients >= 75 years
  Arms: Prasugrel

SUMMARY:
Clopidogrel low response is associated with a significantly higher risk for ischemic complications after percutaneous coronary intervention. Ticagrelor and prasugrel are more potent platelet inhibitory drugs and both have been shown to significantly reduce ischemic events as compared to clopidogrel. No direct comparison between ticagrelor and prasugrel in terms of their antiplatelet efficacy exists. The aim of this study is to assess the antiplatelet treatment efficacy of ticagrelor versus prasugrel over time in confirmed clopidogrel low responders undergoing percutaneous coronary intervention.

ELIGIBILITY:
Inclusion Criteria:

* successful PCI
* 600 mg clopidogrel pretreatment
* clopidogrel low response assessed with electrode aggregometry (>= 486 AU*min)
* written informed consent

Exclusion Criteria:

* Contraindications or allergies against study drugs
* Anemia
* Any surgery < 6 weeks
* Increased bleeding risk
* Oral anticoagulation
* platelet count < 100.000/µl
* Prior history of stroke or pathologic intracranial findings
* GPIIb/IIIa antagonists < 10 days or periprocedural
* Age > 80 years, < 18 years
* Body weight < 60 kg
* Cardiogenic shock
* Increased risk of bradycardia
* Moderate liver disease
* Kidney dialysis
* Intake of CYP 3A4 inhibitors
* Pregnancy or lactation
* Missing pregnancy test for women capable of bearing children

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2011-09; Primary Completion 2014-04 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
ADP-induced platelet aggregation after randomized treatment with ticagrelor or prasugrel | Day 2 post randomization

SECONDARY OUTCOMES:
Proportion of low responders in ticagrelor or prasugrel group | Day 2 post randomization
  Low platelet response is defined as platelet aggregation values >=468 AU*min
Proportion of enhanced responders in ticagrelor or prasugrel group | Day 2 post randomization
  Enhanced platelet response is defined as platelet aggregation values <= 188 AU*min

CONTACTS AND LOCATIONS:
Overall Officials: Katharina Mayer, MD, Principal Investigator — Deutsches Herzzentrum München; Martin Orban, MD, Principal Investigator — Klinikum der Ludwig-Maximilian-Universität München, Campus Großhadern; Daniel Aradi, MD, Principal Investigator — Heart Center Balatonfüred, Dept. of Cardiology
Locations (3):
- Germany (2):
  - Deutsches Herzzentrum, München, Bavaria
  - Klinikum der Ludwig-Maximilians-Universität München, München, Bavaria
- Heart Center Balatonfüred, Dept. of Cardiology, Balatonfüred, Hungary

REFERENCES:
- [Background] Sibbing D, Braun S, Morath T, Mehilli J, Vogt W, Schomig A, Kastrati A, von Beckerath N. Platelet reactivity after clopidogrel treatment assessed with point-of-care analysis and early drug-eluting stent thrombosis. J Am Coll Cardiol. 2009 Mar 10;53(10):849-56. doi: 10.1016/j.jacc.2008.11.030. PMID 19264241
- [Background] Wiviott SD, Braunwald E, McCabe CH, Montalescot G, Ruzyllo W, Gottlieb S, Neumann FJ, Ardissino D, De Servi S, Murphy SA, Riesmeyer J, Weerakkody G, Gibson CM, Antman EM; TRITON-TIMI 38 Investigators. Prasugrel versus clopidogrel in patients with acute coronary syndromes. N Engl J Med. 2007 Nov 15;357(20):2001-15. doi: 10.1056/NEJMoa0706482. Epub 2007 Nov 4. PMID 17982182
- [Background] Wallentin L, Becker RC, Budaj A, Cannon CP, Emanuelsson H, Held C, Horrow J, Husted S, James S, Katus H, Mahaffey KW, Scirica BM, Skene A, Steg PG, Storey RF, Harrington RA; PLATO Investigators; Freij A, Thorsen M. Ticagrelor versus clopidogrel in patients with acute coronary syndromes. N Engl J Med. 2009 Sep 10;361(11):1045-57. doi: 10.1056/NEJMoa0904327. Epub 2009 Aug 30. PMID 19717846